CLINICAL TRIAL: NCT06682572
Title: A Phase 2 Study of Avutometinib (VS-6766, a Dual RAF/MEK Inhibitor) In Combination With Defactinib (FAK Inhibitor) in Recurrent Low-Grade Serous Ovarian Cancer (LGSOC) in Japanese Patients
Brief Title: A Study of Avutometinib + Defactinib in Recurrent Low-Grade Serous Ovarian Cancer in Japanese Patients
Acronym: RAMP201J
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Collaborators: Japanese Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-201J; jRCT2021240021 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Serous Ovarian Cancer; Ovarian Cancer
Keywords: KRAS; KRAS wt; KRAS mt
MeSH Terms: conditions — Ovarian Neoplasms | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- avutometinib + defactinib (Experimental): Avutometinib 3.2mg, PO, twice weekly for 21 days on, 7 days off in a 28-day (4 weeks) cycle in combination with defactinib 200 mg, PO, twice daily for 21 days on, 7 days off in a 28-day (4 week) cycle.
  Interventions: Drug: Avutometinib (VS-6766) + Defactinib (VS-6063)

INTERVENTIONS:
Drug: Avutometinib (VS-6766) + Defactinib (VS-6063) — combination therapy

SUMMARY:
This study will confirm the safety and efficacy of avutometinib in combination with defactinib in Japanese patients with recurrent Low-Grade Serous Ovarian Cancer (LGSOC)

DETAILED DESCRIPTION:
This is a multi-center, open label Phase 2 study designed to evaluate safety and tolerability and confirm efficacy by BICR of avutometinib in combination with defactinib in Japanese patients with molecularly profiled recurrent LGSOC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven LGSOC (ovarian, peritoneal)
* Documented mutational status of KRAS by validated diagnostic test of tumor tissue
* Documented disease progression (radiographic or clinical) or recurrence of LGSOC and have received at least one platinum-based chemotherapy agent
* Measurable disease according to RECIST 1.1
* An Eastern Cooperative Group (ECOG) performance status ≤ 1.
* Adequate organ function
* Adequate recovery from toxicities related to prior treatments
* Agreement to use highly effective method of contraceptive, if necessary

Exclusion Criteria:

* Systemic anti-cancer therapy within 4 weeks of the first dose of study therapy
* Co-existing high-grade ovarian cancer or another histology
* History of prior malignancy, excluding ovarian cancer, with recurrence <3 years from the time of enrollment
* Major surgery within 4 weeks
* Symptomatic brain metastases requiring steroids or other interventions
* Known SARS-Cov2 infection (clinical symptoms) ≤28 days prior to first dose of study therapy
* For subjects with prior MEK exposure, Grade 4 toxicity deemed related to the MEK inhibitor
* Active skin disorder that has required systemic therapy within the past year
* History of rhabdomyolysis
* Concurrent ocular disorders
* Concurrent heart disease or severe obstructive pulmonary disease
* Patients with the inability to swallow oral medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall response rate (ORR; partial response [PR] + complete response [CR] | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate (ORR; partial response [PR] + complete response [CR] defined according to Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) as assessed by the blinded independent central radiology review committee (BICR)

SECONDARY OUTCOMES:
Duration of Response | 12 months
  From the time of first dose of study intervention to PD as assessed by RECIST 1.1 or death from any cause
Objective response rate (ORR) | 12 months
  From the time of first dose of study intervention to PD as assessed by RECIST 1.1 by Investigator or death from any cause.
Progression free survival (PFS) | 24 months
  From the time of first dose of study intervention to first documentation of progressive disease (PD) or death by any cause
Disease control rate (DCR) | 6 months
  CR + PR + SD
Clinical benefit rate | 6 months
  CR + PR + (SD >6 months)
Overall Survival (OS) | up to 2 years
  From the time of first dose of study intervention to PD as assessed by RECIST 1.1 or death from any cause
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 18 months
  Count of AE and SAEs by grade, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale
Area under the plasma concentration-time curve (AUC) of avutometinib, defactinib and relative metabolites | 9 months
  Area under Plasma Concentration (AUC) 0 to t
Maximum plasma concentration (Cmax) of avutometinib, defactinib and relative metabolites | 9 months
  Maximum Plasma Concentration

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume, Fukuoka
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Jikei University Hospital, Minato, Tokyo

IPD SHARING:
Plan to Share IPD: No